CLINICAL TRIAL: NCT04108338
Title: Prospective Comparisons of Survival Outcomes, Safety Profile, and Probability of Returning to Society Between Three Randomized Controlled Trials and Real-world Evidence in Nasopharyngeal Carcinoma.
Brief Title: Prospective Comparisons of Clinical Trial and Real-world Outcomes in Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Other Study IDs: 2019-FXY-239
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Clinical trial; Real-world study; Nasopharyngeal carcinoma; Pragmatism; Survival; Return to society
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CCRT-randomized clinical trial: Trial patients receiving CCRT
  Interventions: Other: Trial setting
- CCRT-real-world database: Patients receiving CCRT from real-world database
- IC+CCRT-randomized clinical trial: Trial patients receiving IC+CCRT
  Interventions: Other: Trial setting
- IC+CCRT-real-world database: Patients receiving IC+CCRT from real-world database

INTERVENTIONS:
Other: Trial setting — Study results from clinical trials usually have been found not work efficiently in clinical practice. This outcome disparity may be caused by different pragmatic features of medical environment, also known as study setting such as trial setting and real-world setting, in which biases inherent to clinical trial design restrict its applicability even though all confounding factors are avoided.
  Other Names: Explanatory medical environment; Non-pragmatic features
  Groups: CCRT-randomized clinical trial; IC+CCRT-randomized clinical trial

SUMMARY:
Study results from randomized controlled trials (RCTs) usually have been found not adequately inform practice. A RCT is optimized to determine efficacy, while real-world study is conducted in a routine care setting aimed to determine effectiveness. Thus, it is necessary to evaluate the pragmatism of clinical trials for a better understanding of the external generalizability. Nonetheless, comparative pragmatic features of RCTs and real-world studies still lack well elucidation. By capitalizing on a nasopharyngeal carcinoma (NPC)-specific big-data, real-world database and individual patient data extracted from three landmark RCTs, investigators conducted the direct comparison of NPC cohorts receiving same treatment strategy in clinical trial versus real-world settings, and examined the comparative pragmatic features and their influences on survival outcomes, safety profile, and the probability of returning to society.

DETAILED DESCRIPTION:
Study results from randomized controlled trials (RCTs) usually have been found not adequately inform practice. A RCT is optimized to determine efficacy. Such trials were performed with relatively small samples at sites with experienced investigators and highly selected participants, they could be overestimating benefits and underestimating harm. Real-world study is conducted in a routine care setting aimed to determine effectiveness. Thus, it is necessary to evaluate the pragmatism of clinical trials for a better understanding of the external generalizability. Nonetheless, comparative pragmatic features of RCTs and real-world studies still lack well elucidation. Nasopharyngeal carcinoma (NPC) is a malignant head and neck cancer with the highest incidences in endemic regions such as Southern China, where over 60,600 new cases were diagnosed in 2015 representing 40% of all cases worldwide. Studies conducted in China are critical in optimizing clinical decision-making of NPC. In the past two decades, the recommendation level of induction chemotherapy (IC) + concurrent chemoradiotherapy (CCRT) has been improved evidently from Category 3 to 2A, and CCRT alone has long been a stable (Category 2B) and classic treatment option of NPC and therefore becomes the most commonly used control group in comparative studies. By capitalizing on a NPC-specific big-data, real-world database via a cancer registry in Southern China and individual patient data extracted from the three landmark RCTs, investigators conducted the direct comparison on IC+CCRT cohort or CCRT cohort of clinical trial versus real-world settings, and examined the comparative pragmatic features and their influences on survival outcomes, safety profile, and the probability of returning to society, with the aim to provide new insight into the optimization of trial design and the translation of study evidences into tangible benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated in our center from April 2009 to December 2016;
2. All patients were pathologically diagnosed, non-metastatic nasopharyngeal carcinoma;
3. Only included cases staged as T3-4N1 & T1-4N2-3 according to the 6th or 7th edition American Joint Committee on Cancer / Union for International Cancer Control (AJCC/UICC) system;
4. For trial patients, treatment strategies only limited to concurrent chemoradiotherapy, induction chemotherapy combined with concurrent chemoradiotherapy, or concurrent chemoradiotherapy combined with adjuvant chemotherapy;
5. For patients from real-world database, patients are permitted to receive additional targeted therapy to standard chemoradiotherapy, as far as it met clinical needs and was approved by physicians.
6. The patient's basic information, prognosis related data, and follow-up data are complete.

Exclusion Criteria:

1. The clinical stage of T3-4N0 was excluded;
2. Cases from large real-world databases need to exclude patients who participate in clinical trials;

Ages: 8 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locoregionally advanced nasopharyngeal carcinoma (T3-4N1 and T1-4N2-3). There are two parts of the constitution of study population.
  Part 1. 1,468 subjects from three phase 3 randomized controlled trials ((NCT00677118, NCT01245959, and NCT01872962) that were conducted by our research team and had been published.
  Part 2. 3,980 subjects from the NPC-specific big-data, real-world database via a cancer registry in Southern China.
Sampling Method: Non-Probability Sample
Enrollment: 5448 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5-year
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive.
Failure-free survival (FFS) | 5-year
  Failure-free survival is measured from day of diagnosis to locoregional failure, distant failure, or death from any cause, whichever occurred first.
Locoregional failure-free survival (LRFFS) | 5-year
  Locoregional failure-free survival is measured from day of diagnosis to first locoregional failure.
Distant failure-free survival (DFFS) | 5-year
  Distant failure-free survival is measured from day of diagnosis to distant failure.
Probability of studying/work stoppage caused by disease and treatment | 5-year
  Probability of learning (students who are in college/university/school before illness) or work (staff who are working before illness) stoppage due to illness and treatment.
Probability of returning to studying/work after suspending | 5-year
  Probability of returning to learning (students who are in college/university/school before illness) or work (staff who are working before illness) after suspending due to illness and treatment.

SECONDARY OUTCOMES:
Incidence of radioactive brain injury | 5-year
  Incidence of radioactive brain injury according to the Common Terminology Criteria for Adverse Events (version 4.0).
Incidence of hearing loss | 5-year
  Incidence of hearing loss according to the Common Terminology Criteria for Adverse Events (version 4.0).
Incidence of blind | 5-year
  Incidence of blind according to the Common Terminology Criteria for Adverse Events (version 4.0).
Incidence of decreased taste | 5-year
  Incidence of decreased taste according to the Common Terminology Criteria for Adverse Events (version 4.0).
Incidence of second cancer | 5-year
  Incidence of second cancer according to the Common Terminology Criteria for Adverse Events (version 4.0).
Incidence of dysphagia | 5-year
  Incidence of dysphagia according to the Common Terminology Criteria for Adverse Events (version 4.0).
Incidence of malnutrition | 5-year
  Incidence of malnutrition according to the Common Terminology Criteria for Adverse Events (version 4.0).
Incidence of hypothyroidism | 5-year
  Incidence of hypothyroidism according to the Common Terminology Criteria for Adverse Events (version 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Booth CM, Tannock IF. Randomised controlled trials and population-based observational research: partners in the evolution of medical evidence. Br J Cancer. 2014 Feb 4;110(3):551-5. doi: 10.1038/bjc.2013.725. Epub 2014 Jan 14. No abstract available. PMID 24495873
- [Background] Prince RM, Atenafu EG, Krzyzanowska MK. Hospitalizations During Systemic Therapy for Metastatic Lung Cancer: A Systematic Review of Real World vs Clinical Trial Outcomes. JAMA Oncol. 2015 Dec;1(9):1333-9. doi: 10.1001/jamaoncol.2015.3440. PMID 26378774